CLINICAL TRIAL: NCT02491034
Title: DESEO: DEpression Screening and Education: Options to Reduce Barriers to Treatment
Acronym: DESEO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Arlington (Other)
Collaborators: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2015-0336
Record Dates: First submitted 2015-07-02; First posted 2015-07-07 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Depression
Keywords: Depression; Hispanics; Stigma; Barriers to Treatment
MeSH Terms: conditions — Depression; Social Stigma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): Depression Education Intervention
  Interventions: Behavioral: Depression Education Intervention

INTERVENTIONS:
Behavioral: Depression Education Intervention — Depression Education Intervention (DEI) designed to increase disease literacy, and dispel myths about depression and its treatment among Hispanic patients thus reducing stigma and increasing treatment engagement.

SUMMARY:
The purpose of this project is to implement a Depression Education Intervention (DEI) designed to increase disease literacy, and dispel myths about depression and its treatment among Hispanic patients thus reducing stigma and increasing treatment engagement. This project will be conducted at one community health center whose patient population is majority Hispanic.

DETAILED DESCRIPTION:
Barriers to depression treatment among Hispanic populations include persistent stigma, inadequate doctor patient communication (DPC) and resultant sub-optimal use of anti-depressant medications. Stigma is primarily perpetuated due to inadequate disease literacy and cultural factors. Common concerns about depression treatments among Hispanics include fears about the addictive and harmful properties of antidepressants, worries about taking too many pills, and the stigma attached to taking psychotropic medications.

Primary care settings often are the gateway to identifying undiagnosed or untreated mental health disorders, particularly for people with comorbid physical health conditions. Hispanics, in particular, are more likely to receive mental health care in primary care settings. Recent recommendations from the U.S. Preventive Services Task Force are that primary care providers screen adult patients for depression only if systems are in place to ensure adequate treatment and follow-up.

Project Purpose, Goals and Objectives Purpose: The purpose of this project is to implement a Depression Education Intervention (DEI) designed to increase disease literacy, and dispel myths about depression and its treatment among Hispanic patients thus reducing stigma and increasing treatment engagement. This project will be conducted at one community health center whose patient population is majority Hispanic.

Goal #1: Patients who screen positive for depression will engage in the Depression Education Intervention (DEI) (two sessions) with a trained Depression Educator.

Objectives:

1. To increase knowledge of depression (signs/symptoms, causes, risk factors, treatment, cultural beliefs, and its role in chronic disease) among Hispanics in a primary care setting as measured by changes in scores from pre- to post- DEI on the Knowledge of Depression-MCQ scale.
2. To reduce perceived cultural stigma about depression and its treatment through a culturally and linguistically appropriate educational intervention as measured by changes in scores from pre- to post- DEI on the Stigma Checklist for Latinos in Primary Care.
3. To increase engagement in depression treatment in primary care by Hispanic patients as measured by the iPad Depression Screening application, which will record the treatment decision after the diagnosis and measure the number of patients engaged in depression treatment of any kind (pharmacotherapy, counseling, other behavioral intervention) at the time of the DEI and one month after completion of the DEI.

Goal #2: In order to identify patients with depression, all adult primary care patients will be screened for depression utilizing the 9-item Patient Health Questionnaire (PHQ-9) via the iPad Depression Screening application.

Objectives:

1. To systematically screen all adult primary care patients with an iPad Depression Screening application as measured by number of patients screened compared to the number eligible for screening.
2. To increase provider detection of depression in patients through the proper use and interpretation of the PHQ-9 as measured by depression diagnoses recorded in the EHR.

ELIGIBILITY:
Inclusion Criteria:

Adult primary care patients

Exclusion Criteria:

* previous diagnosis of depression and currently in treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
The number of Hispanic patients diagnosed with depression who went on to begin depression treatment. | One month post DEI

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Sanchez, PhD, Principal Investigator — The University of Texas at Arlington

REFERENCES:
- [Derived] Sanchez K, Killian MO, Eghaneyan BH, Cabassa LJ, Trivedi MH. Culturally adapted depression education and engagement in treatment among Hispanics in primary care: outcomes from a pilot feasibility study. BMC Fam Pract. 2019 Oct 21;20(1):140. doi: 10.1186/s12875-019-1031-7. PMID 31638915
- [Derived] Lopez V, Sanchez K, Killian MO, Eghaneyan BH. Depression screening and education: an examination of mental health literacy and stigma in a sample of Hispanic women. BMC Public Health. 2018 May 22;18(1):646. doi: 10.1186/s12889-018-5516-4. PMID 29788998
- [Derived] Sanchez K, Eghaneyan BH, Trivedi MH. Depression Screening and Education: Options to Reduce Barriers to Treatment (DESEO): protocol for an educational intervention study. BMC Health Serv Res. 2016 Jul 29;16:322. doi: 10.1186/s12913-016-1575-3. PMID 27473569